CLINICAL TRIAL: NCT03824613
Title: Urinary microRNA Expression in Endometrial Cancer Patients - a Feasibility Study
Brief Title: Urinary miRNA in Endometrial Cancer Study
Status: Completed | Type: Observational
Sponsor: Royal Cornwall Hospitals Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 2018.RCHT.97.
Record Dates: First submitted 2018-12-05; First posted 2019-01-31 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — miRNA in urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endometrial cancer patients
  Interventions: Diagnostic Test: Urinary miRNA
- Control group: Patients without cancer
  Interventions: Diagnostic Test: Urinary miRNA

INTERVENTIONS:
Diagnostic Test: Urinary miRNA — MiRNA detection in urine

SUMMARY:
This study is a prospective feasibility study with the addition of a retrospective cohort study on the the expression of microRNA in urine in endometrial cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of endometrial cancer
* Age: 18 years or older

Exclusion Criteria:

* Prior or coexisting other malignancies
* Autoimmune disorders (other than diabetes mellitus)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Endometrial cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2020-03-26 (Actual); Study Completion 2020-03-26 (Actual)

PRIMARY OUTCOMES:
Accuracy of predictive value of miRNA test in detecting endometrial cancer | 6 months
  To determine if miRNA can distinguish endometrial cancer patients from healthy patients

SECONDARY OUTCOMES:
Correlation to final histology | 6 months
  To determine how well miRNA correlates with final histology, i.e. can miRNA determine the subtype of endometrial cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Cornwall Hospital, Truro, Cornwal, United Kingdom

IPD SHARING:
Plan to Share IPD: No